CLINICAL TRIAL: NCT06708208
Title: Voluntary Termination and Medical Termination of Pregnancy for Maternal, Psychological or Social Reasons At Women's Center ( La Maison Des Femmes) in Saint-Denis
Brief Title: Requests for Voluntary Termination and Medical Termination of Pregnancy for Maternal, Psychological or Social Reasons At the Women's Center ( La Maison Des Femmes) in Saint-Denis :
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0057_MATER_28bis
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Pregnancy; Violence Against Women (VAW); Violence; Abortion; Termination of Pregnancy; Voluntary Termination of Pregnancy; Medical Abortion
Keywords: pregnancy; voluntary termination of pregnancy; violence; abortion; termination of pregnancy; medical abortion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In France, Article L2213-1 of the Public Health Code (law of July 4, 2001) clearly establishes that "voluntary termination of pregnancy may be performed at any time if two doctors, who are part of a multidisciplinary team, certify-after this team has provided its advisory opinion-that continuing the pregnancy seriously endangers the woman's health." Consequently, when a request for termination of pregnancy is made within the first sixteen weeks of amenorrhea, patients exercise complete autonomy in their decision-making. This process is unequivocally recognized as voluntary termination of pregnancy (VTP).

If an abortion is performed after the pregnancy has ended, the patient's request must undergo a multidisciplinary assessment. This procedure is known as medical termination of pregnancy for maternal indications.

There are generally two categories of indications for this procedure:

Organic reasons such as progressive cancer or severe heart disease. Psychosocial reasons: which include psychological and social factors.

In the case of medical terminations of pregnancy for psychological or social reasons, the National College of French Gynaecologists and Obstetricians (CNGOF) recommends that these requests be formally documented within the centers where patients receive care. However, there is considerable variability in how these practices are implemented across different locations. Furthermore, the existing literature reveals a significant lack of epidemiological and clinical data on the subject, highlighting the need for more comprehensive research in this area.

Opened in 2016, the Maison des Femmes (Women's Center) in Saint-Denis houses a family planning center and a multi-professional support service for patients who have experienced violence. It provides care for many women who have sought a termination of pregnancy but have exceeded the legal time limit for abortion.

A study conducted in 2021-2022, as part of a medical thesis, revealed a significantly high prevalence of violence experienced by women seeking a pregnancy termination for non-medical reasons at Delafontaine Hospital. The findings indicated that 65% of these patients had suffered from violence.

To strengthen our epidemiological findings, we propose a study comparing this group of women with another group who had an abortion during the same timeframe.

ELIGIBILITY:
Inclusion Criteria:

* Patients (minors or adults) who have been seen at the Women's center (Maison des Femmes) for assistance with a request of termination of pregnancy for maternal, psychological and/or social reasons, including patients under legal protection (guardianship, curatorship) at the time of the consultation.
* medical consultation between 01/01/2016 and 28/02/2022.

Exclusion Criteria:

* Refusal of participation (patient or guardian)
* Opposition to the use of data

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women who are pregnant.
Study Population: Patients who expressed a request for an IMG for non-somatic maternal reasons
Sampling Method: Non-Probability Sample
Enrollment: 107 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Demographic data | 1 day
  Age
Demographic data | 1 day
  Birth place
Demographic data | 1 day
  Migration history
Medical history | 1 day
  Term of abotion
Violence's history | 1 day
  Description of the violence. Current situation of violence.

CONTACTS AND LOCATIONS:
Locations (1):
- Maison des femmes, Saint-Denis, Seine saint denis, France

IPD SHARING:
Plan to Share IPD: No